CLINICAL TRIAL: NCT06274606
Title: Exercise Training Study Before Bariatric Surgery
Acronym: BaSE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Project during development was discontinued before the enrollment of participants
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Damon Swift, Associate Professor, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HSR230106
Record Dates: First submitted 2024-01-18; First posted 2024-02-23 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Bariatric Surgery Candidate
Keywords: Bariatric surgery; Obesity; Insulin sensitivity; Exercise intervention
MeSH Terms: conditions — Obesity; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: In accordance with a parallel study design, 30 pre-bariatric-surgery patients will be randomized in a 1:1 ratio to either undergo 8-weeks of pre-operative standard of care or 8-weeks of pre-operative standard of care plus moderate exercise prior to undergoing bariatric-surgery. Randomization scheme: The randomization will be generated utilizing a permuted block randomization scheme in which 5 blocks of 6 treatment assignments (3 per treatment) will be generated via a computer algorithm. The 6 treatment assignments of each block will be listed in random sequential order and the treatment assignments will be assigned according to the random sequential order. The randomization will be generated by our biostatistician.
Masking Description: Randomization will be completely random and will only be known by biostatistician and study coordinator in department but not on study to retain true randomization unaffected by study team.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise Group (EX-group) (Experimental): The EX-group will complete 8 weeks of supervised aerobic exercise training. The EX-group will also continue normal care with bariatric doctors and nurses along with the exercise intervention.
  Interventions: Other: Exercise Group
- Standard Care Only Group (SC-group) (No Intervention): The SC-group will only complete the orientation visit and testing visits. The participants that are randomized to this group will continue normal care with bariatric doctors and nurses. They will participate in study assessment visits only.

INTERVENTIONS:
Other: Exercise Group — Previously sedentary adults awaiting bariatric surgery will be randomized to either an Exercise group (EX-group) or Standard care only group (SC-group) for 8 weeks. Outcome visits will occur before the exercise intervention, after the exercise intervention, and after surgery
  Arms: Exercise Group (EX-group)

SUMMARY:
The goal of this clinical trial is to figure out if 8 weeks of walking exercise before bariatric surgery improves risk factors for diabetes and other markers of health. This is important as it may help reduce complications after surgery, improve health markers and increase physical activity levels after surgery (which is an important marker of maintaining bariatric weight loss). The main question that this study is trying to answer is whether walking improves a risk factor for type 2 diabetes called insulin sensitivity (how well your body is able to use glucose).

Adults planning to have bariatric surgery will be recruited from the Charlottesville VA area. Before they have their surgery, participants will be randomly assigned (like flipping a coin) to a group that participates in 8 weeks of walking on a treadmill (2-3 times a week) or a group that does their normal care before bariatric surgery.

Researchers will compare the effects of walking before bariatric surgery on:

* Insulin sensitivity (diabetes risk factor)
* Health of blood vessels
* Rate of complications after surgery
* Weight
* Body Fat
* Fitness level

DETAILED DESCRIPTION:
The purpose of the present study is to evaluate the impact of 8 weeks of supervised aerobic exercise prior to bariatric surgery on insulin sensitivity using the hyperinsulinemic-euglycemic clamp. Participants will be recruited from the area surrounding the UVA hospital, while the primary outcome will be insulin sensitivity as measured by the hyperinsulinemic-euglycemic clamp procedure and secondary outcomes include the effects of the exercise intervention on surgical outcomes and cardiometabolic and arterial health in bariatric patients.

Objectives:

Primary Objective: To investigate the effects of exercise + standard care and standard care only in obese individuals prior to bariatric surgery on insulin sensitivity after bariatric surgery.

Secondary Objectives: To examine the effects of exercise + standard care and standard care only in obese individuals prior to bariatric surgery on surgical outcomes, such as length of stay post-surgery, and other clinically relevant outcomes, such as cardiometabolic and arterial health, in adults following bariatric surgery.

Hypotheses:

Primary Hypothesis: An 8-week exercise intervention before bariatric surgery will improve insulin sensitivity as measured by the hyperinsulinemic-euglycemic clamp following bariatric surgery.

Secondary Hypothesis: An 8-week exercise intervention will improve clinically relevant post-surgical outcomes, such as surgical outcomes, quality of life, arterial health, and other cardiometabolic factors following bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* BMI: 35 - 45 kg/m2. For adults of Asian race or descent, the BMI cutoff is between 25-27.5 kg/m2 to be considered for surgery and thus will be considered for inclusion in this study.
* Considered sedentary based on self-reported inactivity of < 2-3 x/week of MVPA within previous 3 months before enrollment.
* Able to walk without use of assistive device, such as cane or walker for ≥ 10 minutes.
* Surgery approved within 6-9 months of initial visit.
* Signed approval from study physician (Dr. Catherine W. Varney; Medical PI of study) that participant is capable to participate.
* Willingness to accept group randomization assignment.

Exclusion Criteria:

* Any serious medical conditions, such as cancer; history cardiovascular disease of stroke, heart attack, or heart failure; type 1 diabetes mellitus; severe psychiatric illness (such as severe depression); kidney disease.
* Autoimmune diseases such as lupus, multiple sclerosis, Graves' disease, or rheumatoid arthritis.
* HIV or tuberculosis.
* Currently taking medications that lead to significant weight loss (e.g., semaglutide; tirzepatide, etc).
* Resting SBP > 150 mmHg, DBP > 100 mmHg.
* Current pregnancy or plans to become pregnant during intervention.
* Plans to be away from the Charlottesville, VA area for > 1 week during intervention or plans of relocating during the intervention.
* Any medical or health condition (e.g., musculoskeletal, orthopedic, or neurological conditions) that is contraindicated for safe exercise testing and training.
* Previous weight-loss surgeries or revisions

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
Insulin sensitivity | Change from baseline to after surgery (12 weeks)
  Insulin sensitivity measured via the hyperinsulinemic-euglycemic clamp

SECONDARY OUTCOMES:
Surgical outcomes - readmission within 30 days of surgery | within 30 days
  Variables recorded after surgery such as readmission within 30 days of surgery
Surgical outcomes - IV treatment as an outpatient | Change from baseline to after surgery (12 weeks)
  Variables recorded after surgery such as IV treatment as an outpatient
Surgical outcomes - emergency department visits | Change from baseline to after surgery (12 weeks)
  Variables recorded after surgery such as emergency department visits
Surgical outcomes - time of surgery | Intraoperative
  Variables recorded after surgery such as time of surgery (min).
Surgical outcomes - length of stay after surgery completion | Change from baseline to after surgery (12 weeks)
  Variables recorded after surgery such as length of stay after surgery
Flow-mediated dilation (FMD) | Change from baseline to after surgery (12 weeks)
  Endothelial function measured via flow mediated dilation (FMD) (%) - indication of shear-stress-mediated dilation following occlusion
Pulse-wave analysis (PWA) | Change from baseline to after surgery (12 weeks)
  Pulse-wave analysis (PWA) as measured with a SphygmoCor Xcel to measure brachial systolic and diastolic pressures and to capture a brachial waveform.
Pulse-wave velocity (PWV) | Change from baseline to after surgery (12 weeks)
  Pulse-wave velocity (PWV) as measured with a SphygmoCor Xcel to measure the blood pressure waveforms at the carotid and femoral artery sites.
Body fat | Change from baseline to after surgery (12 weeks)
  Dual-energy x-ray absorptiometry (DEXA) will be used to access body fat (g)
Lean body mass | Change from baseline to after surgery (12 weeks)
  Dual-energy x-ray absorptiometry (DEXA) will be used to access lean body mass
Bone mineral density | Change from baseline to after surgery (12 weeks)
  Dual-energy x-ray absorptiometry (DEXA) will be used to access bone mineral density (g)
Visceral adiposity | Change from baseline to after surgery (12 weeks)
  Dual-energy x-ray absorptiometry (DEXA) will be used to access visceral adiposity measures (g)
Weight | Change from baseline to after surgery (12 weeks)
  Body weight measured on a level beam scale; minimum value 0 kg-500kg; higher scores tend to suggest worsened outcomes
Blood Lipids | Change from baseline to after surgery (12 weeks)
  Cholesterol values, including HDL-C, LDL-C, and VLDL-C (mg/dL) from intravenous line
Plasma glucose | Change from baseline to after surgery (12 weeks)
  Plasma glucose (mg/dL) from intravenous line
Plasma insulin | Change from baseline to after surgery (12 weeks)
  Plasma insulin (uIU/dL) from intravenous line
Hemoglobin A1c | up to 12 weeks
  Hemoglobin A1C (%) - an average of blood glucose levels in the previous 3 months
Cardiorespiratory fitness | Change from baseline to after surgery (12 weeks)
  Vo2 max measured via a maximal exercise test on a treadmill
Quality of life (SF-36) | Change from baseline to after surgery (12 weeks)
  Quality of life will be assessed via the SF-36 and the variables included in the questionnaire are physical functioning (PF), role physical (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role emotional (RE), and mental health (MH)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Within 1 year of study completion
Access Criteria: Access to UVA Health portals, including UVA Health REDCap